CLINICAL TRIAL: NCT01750073
Title: A Phase II Study of Neoadjuvant Chemotherapy With and Without Trastuzumab in Patients With Breast Cancer
Brief Title: Paclitaxel & Cyclophosphamide With or Without Trastuzumab Before Surgery in Treating Previously Untreated Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0264-12-FB; NCI-2012-01372 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2023-12-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Estrogen Receptor Negative; Estrogen Receptor Positive; HER2/Neu Negative; HER2/Neu Positive; Invasive Breast Carcinoma; Progesterone Receptor Negative; Progesterone Receptor Positive; Stage IA Breast Cancer; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel; Taxes; Radiotherapy; Radiation; Trastuzumab; PF-05280014

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (chemotherapy, surgery, post-operative therapy) (Experimental): See Detailed Description
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery; Biological: Trastuzumab

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo mastectomy or breast conserving surgery
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar PF-05280014

SUMMARY:
This phase II trial studies the side effects and how well giving paclitaxel and cyclophosphamide with or without trastuzumab before surgery works in treating patients with previously untreated breast cancer. Drugs used in chemotherapy, such as paclitaxel and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, may block tumor growth in different ways by targeting certain cells. Giving combination chemotherapy with or without trastuzumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicities and tolerability of a neoadjuvant dose-dense regimen cyclophosphamide and paclitaxel with or without trastuzumab/radiation therapy (as clinically indicated) in patients with newly diagnosed stage T1cN0 and II-III breast cancer; followed by maintenance trastuzumab in human epidermal growth factor receptor 2 (HER2) positive OR adriamycin (doxorubicin hydrochloride) followed by radiation therapy (RT) in stage II-III triple negative HER2 (-), estrogen receptor (ER) (-), progesterone receptor (PR) (-) stage T1cN0 and II-III breast cancer patients.

II. To determine the pathological complete response rate (pCR) of this treatment regimen.

III. To identify possible gene expression profile signatures from whole genome array analysis that correlate with clinical response/resistance to chemotherapy as measured by pathologic complete response rate (pCR).

OUTLINE:

NEOADJUVANT THERAPY: Patients receive paclitaxel intravenously (IV) over 3 hours and cyclophosphamide IV over 1 hour on day 1. Patients with HER2-positive cancer also receive trastuzumab IV over 30 minutes on day 1. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients without metastasis undergo mastectomy or breast conserving surgery 4-8 weeks later.

POST-SURGERY/SYSTEMIC THERAPY:

HER2-POSITIVE PATIENTS: Patients receive standard radiation therapy. Patients also receive trastuzumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

ER/PR POSITIVE PATIENTS: Patients receive standard adjuvant hormonal or endocrine therapy.

STAGE T1cN0 TRIPLE NEGATIVE PATIENTS: Patients receive standard radiation therapy.

STAGE II-III TRIPLE NEGATIVE PATIENTS: Patients receive doxorubicin hydrochloride IV over 15 minutes on day 1. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients also receive standard radiation therapy.

After completion of study treatment, patients are followed up every 3 months for 2 years, and then annually thereafter for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically proven invasive breast cancer without distant metastases; a clinical tumor classification of tumor size must be at least 1 cm with or without clinical pathologic evidence of positive nodes
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* At least one lesion that can be accurately measured in two dimensions utilizing mammogram, ultrasound, or magnetic resonance imaging (MRI) images to define specific size and validate complete clinical and pathologic response
* Patients who received radiation therapy > 5 years ago for malignancies other than breast cancer and whose radiation therapy field is not overlapping with the 20% isodose line of current radiation field are eligible, provided that radiation therapy was completed > 5 years ago and that there is no evidence of the second malignancy at the time of study entry
* Absolute neutrophil count greater than or equal to 1,500/mcl
* Platelet count equal to or greater than 150,000/mcl
* Alkaline phosphatase equal or less than 1.5 times the upper limit of normal (ULN)
* Total bilirubin equal to or less than 1.5 times the ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) no greater than 1.5 times the ULN
* Creatinine less than 1.5 times the ULN
* All included patients must have normal cardiac function as defined by an ejection fraction of >= 50% and no decrease in wall motion by echocardiogram
* The patient must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts
* Women of reproductive potential must be non-pregnant and non-nursing and must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following treatment
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiating study; (no childbearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)

Exclusion Criteria:

* Any patient with inflammatory breast cancer or stage IV or confirmed metastatic disease
* Patients who have had any prior chemotherapy, or endocrine therapy for the treatment of breast cancer or any other cancer
* Patients who cannot undergo surgery
* Patients with a known or documented anaphylactic reaction or allergy to any of chemotherapy agents used in this protocol, or to antiemetics appropriate for administration in conjunction with protocol-directed therapy
* Uncontrolled inter-current illness including, but not limited to ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, or serious, uncontrolled cardiac arrhythmia, that might jeopardize the ability of the patient to receive the therapy program outlined in this protocol with reasonable safety
* Patients with preexisting grade II peripheral neuropathy
* Pregnant and nursing women are excluded from this study
* Patients with prior malignancy will be excluded except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas
* Inability to cooperate with treatment protocol
* Patients with known human immunodeficiency virus (HIV) infection, infectious hepatitis, type A, B or C, active hepatitis, or hepatic insufficiency
* Patients may not be receiving or have received any other investigational agents during/or within 1 month prior
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amulya C Yellala, MD, Principal Investigator — University of Nebraska
Locations (4):
- United States (4):
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Nebraska Medicine-Village Pointe Cancer Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 99 subjects were enrolled but 7 were screen fails (after signing consent) so only 92 started.
Period: Overall Study
Arm/Group | Treatment (chemotherapy, surgery, post-operative therapy)
Started | 92
HER2-positive | 19
HER2-negative | 73
Completed | 87
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Surgery, Post-operative Therapy)
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.65 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 89
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 80
  More than one race | 0
  Unknown or Not Reported | 0
Stage of Cancer [Count of Participants; unit: Participants]
  Stage I | 22
  Stage II | 65
  Stage IIIA | 5
Her-2 NEU Status (human epidermal growth factor receptor) [Count of Participants; unit: Participants]
  Negative | 73
  Positive | 19
ER Status [Count of Participants; unit: Participants]
  Negative | 35
  Positive | 57
PR Status (progesterone receptors) [Count of Participants; unit: Participants]
  Negative | 49
  Positive | 43
Triple Negative [Count of Participants; unit: Participants]
  No | 63
  Yes | 29
Treatment [Count of Participants; unit: Participants] — PC = Paclitaxel PCH = Paclitaxel + Cyclophospamide PC + Adriamycin = Paclitaxel + Adriamycin
  Participants
    paclitaxel & cyclophosphamide (PC) + Adriamycin | 17
    paclitaxel & cyclophosphamide (PC) | 56
    paclitaxel, cyclophosphamide & trastuzumab (PCH) | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Incidence of Toxicities, Graded According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Number of participants in each subset (Her2 positive and Her2 negative) who experience at least one adverse event [overall incidence of toxicities, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0].
Time Frame: Up to 30 days after completion of study treatment, maximum of 114 days
Population: All subjects who received at least one cycle of treatment and experienced an adverse event.
Measure: Count of Participants; unit: Participants
Groups:
- Her-2 Negative; Her-2 Positive: See Detailed Description
  Cyclophosphamide: Given IV
  Doxorubicin Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Radiation Therapy: Undergo RT
  Therapeutic Conventional Surgery: Undergo mastectomy or breast conserving surgery
  Trastuzumab: Given IV
Arm/Group | Her-2 Negative | Her-2 Positive
Number analyzed (Participants) | 73 | 19
Participants | 73 | 19

2. Primary Outcome: Overall Severity of Toxicities, Graded According to the NCI CTCAE Version 4.0
Description: Results reported as total events per grade for human epidermal growth factor receptor 2 (HER2)negative and HER2 positive (Overall severity of toxicities, graded according to the NCI CTCAE version 4.0).
Time Frame: Up to 30 days after completion of study treatment, maximum of 114 days
Population: Participant events were analyzed for each group-Her-2 Negative and Her-2 Positive
Measure: Number; unit: Events
Units Other Than Participants: Events
Arm/Group | Her-2 Negative | Her-2 Positive
Number analyzed (Participants) | 73 | 19
Number analyzed (Events) | 1816 | 496
Events
  SAE grade 1 | 1 | 9
  SAE grade 2 | 10 | 4
  SAE grade 3 | 22 | 8
  SAE grade 4 | 2 | 2
  SAE grade 5 | 1 | 1
  Non-SAE grade 1: number analyzed (Events) | 1816 | 302
  Non-SAE grade 1 | 1286 | 302
  Non-SAE grade 2 | 390 | 143
  Non-SAE grade 3 | 93 | 23
  Non-SAE grade 4 | 11 | 4

3. Primary Outcome: Number of Participants in the Subgroups Who Had a Pathologic Complete Response (pCR)
Description: The number of participants in the subgroups who had a pathologic complete response (pCR) determined from the surgical specimen and defined as the absence of invasive carcinoma in both the breast and axilla at microscopic examination of the resection specimen, regardless of the presence of carcinoma in situ.
Time Frame: Up to 12 weeks (after the first 6 courses of treatment), maximum of 168 days
Population: Participants who completed 6 courses of treatment (87). 16 subjects were not evaluated. Total of 71 participants were evaluated.
Measure: Number; unit: participants
Arm/Group | Her-2 Negative | Her-2 Positive
Number analyzed (Participants) | 56 | 15
participants | 13 | 2

4. Secondary Outcome: Clinical Complete Response
Description: The absence of all detectable cancer after treatment is complete.
Time Frame: Up to 2 years
Reporting Status: Not Posted, anticipated posting 2027-06

5. Secondary Outcome: Failure-free Survival (FFS)
Description: The analysis will be based on Kaplan-Meier estimates. FFS will be summarized overall and for human epidermal growth factor receptor 2 (HER2)+ and HER- subsets.
Time Frame: The time from the date of administration of study drug to the date of first appearance of tumor lesions by imaging, or death, assessed up to 2 years
Reporting Status: Not Posted, anticipated posting 2027-06

6. Secondary Outcome: Identification of Gene Expression Profile Signatures That Correlate With Clinical Response as Measured by pCR
Description: The number of the identified mutated genes, the frequency of each gene being validated by reverse transcriptase-polymerase chain reaction (RT-PCR)/Sanger sequencing method, and the functions of these identified genes will be descriptively summarized.
Time Frame: Up to 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival (OAS)
Description: The analysis will be based on Kaplan-Meier estimates. OAS will be summarized overall and for HER+ and HER- subsets.
Time Frame: The time from the date of the date of administration of study drug to the date of death from any cause, assessed up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days after last administration of study medication, maximum of 114 days
Arm/Group | Treatment (chemotherapy, surgery, post-operative therapy)
All-Cause Mortality (participants affected / at risk) | 2/92
Serious Adverse Events (participants affected / at risk) | 16/92
Other Adverse Events (participants affected / at risk) | 92/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (chemotherapy, surgery, post-operative therapy) (N=92)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5
Anemia (Blood and lymphatic system disorders) | 3
Infections and Infestations (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Fever (General disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Neutrophil count decreased (Investigations) | 2
non-cardiac chest pain (General disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Urinary tract infection (Infections and infestations) | 2
white blood cell decreased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Asystole (Cardiac disorders) | 1
Blood bilirubin increased (Investigations) | 1
Cardiac troponin I increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Infusion related reaction (General disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Pericarditis (Cardiac disorders) | 1
Platelet count decreased (Investigations) | 1
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (chemotherapy, surgery, post-operative therapy) (N=92)
Peripheral sensory neuropathy (Nervous system disorders) | 81
Hyperglycemia (Metabolism and nutrition disorders) | 66
Fatigue (General disorders) | 55
Alkaline phosphatase increased (Investigations) | 54
Anemia (Blood and lymphatic system disorders) | 49
Nausea (Gastrointestinal disorders) | 48
Arthralgia (Musculoskeletal and connective tissue disorders) | 41
White blood cell decreased (Investigations) | 38
Myalgia (Musculoskeletal and connective tissue disorders) | 36
Constipation (Gastrointestinal disorders) | 35
Hyponatremia (Metabolism and nutrition disorders) | 35
Headache (Nervous system disorders) | 30
Hypocalcemia (Metabolism and nutrition disorders) | 30
Diarrhea (Gastrointestinal disorders) | 29
Insomnia (Psychiatric disorders) | 29
Bone pain (Musculoskeletal and connective tissue disorders) | 28
Hypokalemia (Metabolism and nutrition disorders) | 26
Alanine aminotransferase increased (Investigations) | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Anxiety (Psychiatric disorders) | 18
Neutrophil count decreased (Investigations) | 17
Pain (General disorders) | 17
Alopecia (Skin and subcutaneous tissue disorders) | 16
Aspartate aminotransferase increased (Investigations) | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Mucositis oral (Gastrointestinal disorders) | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Hypertension (Vascular disorders) | 14
Lymphocyte count decreased (Investigations) | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14
Dysgeusia (Nervous system disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 13
Fever (General disorders) | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13
Platelet count decreased (Investigations) | 13
Creatinine increased (Investigations) | 11
Depression (Psychiatric disorders) | 11
Edema limbs (General disorders) | 11
Hot flashes (Vascular disorders) | 11
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 10
Dizziness (Nervous system disorders) | 10
Flushing (Vascular disorders) | 10
Gastroesophageal reflux disease (Gastrointestinal disorders) | 10
Glucose intolerance (Metabolism and nutrition disorders) | 10
Vomiting (Gastrointestinal disorders) | 9
Blurred vision (Eye disorders) | 8
Dry mouth (Gastrointestinal disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 8
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Upper respiratory infection (Infections and infestations) | 6
Urinary incontinence (Renal and urinary disorders) | 6
Allergic reaction (Immune system disorders) | 5
Palpitations (Cardiac disorders) | 5
Scalp pain (Skin and subcutaneous tissue disorders) | 5
Urinary frequency (Renal and urinary disorders) | 5
Urinary tract infection (Infections and infestations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT01750073/Prot_SAP_000.pdf